CLINICAL TRIAL: NCT02982395
Title: A Phase Ⅲ Study to Evaluate the Efficacy and Safety Of Intravesical Nanoxel®M (Docetaxel-PM) In Bacillius Calmette-Guerin Refractory Non-Muscle Invasive Bladder Cancer
Brief Title: Study to Evaluate the Efficacy and Safety Of Intravesical Nanoxel®M In BCG Refractory NMIBC
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Samyang Biopharmaceuticals Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DPMBLC301
Record Dates: First submitted 2016-11-24; First posted 2016-12-05 (Estimated); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Non Muscle Invasive Bladder Cancer
Keywords: Nanoxel M; Docetaxel PM; Docetaxel; Mitomycin C; BCG; BCG refractory; Non muscle invasive bladder cancer; intravesical; superficial bladder cancer; Urothelial carcinoma; Transitional cell carcinoma
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms; Carcinoma, Transitional Cell | interventions — Polysorbates; Mitomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nanoxel®M (Experimental): 75 mg in 100mL normal saline
  Interventions: Drug: Nanoxel®M
- Mitomycin (Active Comparator): 40 mg in 100mL normal saline
  Interventions: Drug: Mitomycin-C

INTERVENTIONS:
Drug: Nanoxel®M — Intravesical
  Other Names: Polysorbate 80, ethanol free Docetaxel
  Arms: Nanoxel®M
Drug: Mitomycin-C — Intravesical
  Arms: Mitomycin

SUMMARY:
The purpose of this study is to determine whether Nanoxel®M is effective in the treatment of patients with recurrent Ta and T1 who experienced treatment failure with at least one prior BCG intravesical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of superficial transitional cell carcinoma of the bladder (Ta, T1)
* Recurrent superficial bladder cancer refractory to Bacillus Calmette-Guerin (BCG)
* No previous intravesical therapy for 6 weeks
* No history of prior radiation to the pelvis
* Peripheral neuropathy ≤ grade 1
* Eastern Cooperative Oncology Group (ECOG) performance status 0 t0 2
* Adequate hematopoietic and hepatic parameters

Exclusion Criteria:

* Muscle invasive disease (T2-T4)
* Any other malignancy diagnosed within 2 years of study entry (Except basal or squamous cell skin cancers or noninvasive cancer of the cervix)
* Participation in any other research protocol involving administration of an investigational agent within 3 months before study entry
* History of sensitivity reaction to docetaxel
* Prescribed immunosuppressive medications because of a confounding medical condition
* Female patients who were pregnant or lactating

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Recurrence free rate | 1 year
  Recurrence free rate will be summarized as the percentage of participants who achieved a confirmed recurrence free as assessed by urine cytology and cystoscopy. Recurrence means reappearance of high-risk disease (high grade, T1 or CIS) after the start of therapy.

SECONDARY OUTCOMES:
Recurrence free rate | 6 months, 2 years
  Recurrence free rate will be summarized as the percentage of participants who achieved a confirmed recurrence free as assessed by urine cytology and cystoscopy.Recurrence means reappearance of high-risk disease (high grade, T1 or CIS) after the start of therapy.
Overall survival | 2 years
  Time from random assignment to death resulting from any cause.
Number of participants with adverse events as assessed by CTCAE v4.0 | 2 years
  Adverse event (AE) is as any AE occurring or worsening from the first treatment of any study drug to the last dose of the last study drug. Severity grades according to NCI CTCAE version 4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Ja Hyeon Ku, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No